CLINICAL TRIAL: NCT04478305
Title: The Effect of Conjugated Estrogens/ Bazedoxifene (CE/ BZA) on Peri- and Postmenopausal Mood and Anxiety Symptoms: A Pilot Study
Brief Title: Affect of Duavive on Mood & Anxiety Symptoms
Acronym: DOMA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Alison Shea, Menopause and Reproductive Mental Health Specialist, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-7333
Record Dates: First submitted 2020-03-19; First posted 2020-07-20 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Menopause; Depression, Anxiety; Sleep; Menopause Related Conditions
Keywords: hormone replacement therapy
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single group longitudinal study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Other): Patient will be provided with study medication. To be taken once a day for 16 weeks (112 days). Active drug brand name - Duavive/Duavee. Dose consisting of 1 pill of 0.45mg conjugated estrogens and 20mg bazedoxifene as bazedoxifene acetate.
  Interventions: Drug: Duavive 0.45Mg-20Mg Tablet

INTERVENTIONS:
Drug: Duavive 0.45Mg-20Mg Tablet — Duavee, marketed as Duavive in Canada.
  Other Names: Duavive

SUMMARY:
This study evaluates the impact of conjugated estrogens/ bazedoxifene (CE/ BZA) on the mood (depression and anxiety) in peri- and early menopausal women.

DETAILED DESCRIPTION:
During the transition to menopause, women are at risk for developing symptoms of depression and anxiety, and impaired sleep. Fluctuation in estrogen levels appears to play a role in this. The investigators suspect that the administration of estrogens without progesterone, such as conjugated estrogens/ bazedoxifene (CE/ BZA), may improve mood symptoms in this population. In 2017, CE/ BZA was approved for menopausal vasomotor symptoms (VMS) in Canada, but the effect on mood were not examined closely.

The investigators propose a pilot study of 30 peri- and early postmenopausal women, currently seeking treatment for symptoms of depression or anxiety. The participants will go through a round of treatment with CE/BZA. The study will last 16 weeks. The study's objectives are to determine primarily if CE/BZA improves mood among peri- and early postmenopausal women, and secondarily if treatment with CE/BZA improves their sleep.

ELIGIBILITY:
Inclusion Criteria:

* Females between 45-60 years of age
* Able to communicate in English
* In perimenopause as defined by World Health Organization (WHO) Stages of Reproductive Aging Workshop (STRAW) criteria, OR in early menopause (within 10 years of final menstrual period)
* Suffering from Depressive symptoms (10+ on CES-D-10) AND/OR anxiety symptoms (10+ on GAD-7)

Exclusion Criteria:

* Personal history of breast/ ovarian/ endometrial cancer/ endometrial hyperplasia.
* Abnormal uterine bleeding that has not been adequately investigated.
* Active or past venous or arterial thromboembolic disease (deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction, coronary heart disease).
* Active liver disease.
* Known protein C, protein S, or antithrombin deficiency or other known thrombophilic disorders.
* Known or suspected pregnancy, women who may become pregnant, and nursing mothers
* Partial or complete loss of vision due to ophthalmic vascular disease.
* Uncontrolled hypertension (Systolic blood pressure >160mm Hg and/ or diastolic blood pressure >95 mm Hg)
* Endocrine disease (other than thyroid disease) that may adversely affect mood (i.e., Cushing's disease, Addison's disease). For women with abnormal TSH, it will be corrected in advance of trial initiation.
* Active serious suicidal ideation with intent.
* Symptoms of active psychosis.
* Daily use of antidepressive medication.
* Use of other psychoactive or centrally acting medications within 2 weeks before study screening.
* Known hypersensitivity to either CE or BZA.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | At 4 weeks weeks after beginning study
  Assessed by scores on the Center for Epidemiologic Studies Depression Scale (CES-D=10). Any score that is equal to or higher than 10 is considered depressed.
Depressive symptoms | At 8 weeks after beginning study
  Assessed by scores on the Center for Epidemiologic Studies Depression Scale (CES-D). Scores from 0-60, with higher scores indicating higher levels of depression.
Depressive symptoms | At 12 weeks after beginning study
  Assessed by scores on the Center for Epidemiologic Studies Depression Scale (CES-D). Scores from 0-60, with higher scores indicating higher levels of depression.
Depressive symptoms | At 16 weeks after beginning study
  Assessed by scores on the Center for Epidemiologic Studies Depression Scale (CES-D). Scores from 0-60, with higher scores indicating higher levels of depression.
Depressive symptoms | At 4 weeks after beginning study
  Assessed by scores on the Montgomery-Asberg Depression rating Scale (MADRS). The scores range from 0-60, with higher scores indicating higher levels of depression.
Depressive symptoms | At 8 weeks after beginning study
  Assessed by scores on the Montgomery-Asberg Depression rating Scale (MADRS). The scores range from 0-60, with higher scores indicating higher levels of depression.
Depressive symptoms | At 12 weeks after beginning study
  Assessed by scores on the Montgomery-Asberg Depression rating Scale (MADRS). The scores range from 0-60, with higher scores indicating higher levels of depression.
Depressive symptoms | At 16 weeks after beginning study
  Assessed by scores on the Montgomery-Asberg Depression rating Scale (MADRS). The scores range from 0-60, with higher scores indicating higher levels of depression.
Anxiety symptoms | At 4 weeks after beginning study
  Assessed by scores on the Generalized Anxiety Disorder Scale (GAD-7). The scores range from 0-21, with higher scores indicating higher levels of anxiety.
Anxiety symptoms | At 8 weeks after beginning study
  Assessed by scores on the Generalized Anxiety Disorder Scale (GAD-7). The scores range from 0-21, with higher scores indicating higher levels of anxiety.
Anxiety symptoms | At 12 weeks after beginning study
  Assessed by scores on the Generalized Anxiety Disorder Scale (GAD-7). The scores range from 0-21, with higher scores indicating higher levels of anxiety.
Anxiety symptoms | At 16 weeks after beginning study
  Assessed by scores on the Generalized Anxiety Disorder Scale (GAD-7). The scores range from 0-21, with higher scores indicating higher levels of anxiety.

SECONDARY OUTCOMES:
Menopause symptoms | At 4 weeks after beginning study
  Assessed by the Greene Climacteric Scale (GCS). Scores range from 0-21, with higher scores indicating more severe menopausal symptoms.
Menopause symptoms | At 8 weeks after beginning study
  Assessed by the Greene Climacteric Scale (GCS). Scores range from 0-21, with higher scores indicating more severe menopausal symptoms.
Menopause symptoms | At 12 weeks after beginning study
  Assessed by the Greene Climacteric Scale (GCS). Scores range from 0-21, with higher scores indicating more severe menopausal symptoms.
Menopause symptoms | At 16 weeks after beginning study
  Assessed by the Greene Climacteric Scale (GCS). Scores range from 0-21, with higher scores indicating more severe menopausal symptoms.
Total nightly sleep time | At 4 weeks after beginning study
  Assessed by an Actigraph 2 monitor
Total nightly sleep time | At 8 weeks after beginning study
  Assessed by an Actigraph 2 monitor
Total nightly sleep time | At 12 weeks after beginning study
  Assessed by an Actigraph 2 monitor
Total nightly sleep time | At 16 weeks after beginning study
  Assessed by an Actigraph 2 monitor
Sleep onset latency | At 4 weeks after beginning study
  Assessed by an Actigraph 2 monitor
Sleep onset latency | At 8 weeks after beginning study
  Assessed by an Actigraph 2 monitor
Sleep onset latency | At 12 weeks after beginning study
  Assessed by an Actigraph 2 monitor
Sleep onset latency | At 16 weeks after beginning study
  Assessed by an Actigraph 2 monitor
Wake after sleep onset | At 4 weeks after beginning study
  Assessed by an Actigraph 2 monitor
Wake after sleep onset | At 8 weeks after beginning study
  Assessed by an Actigraph 2 monitor
Wake after sleep onset | At 12 weeks after beginning study
  Assessed by an Actigraph 2 monitor
Wake after sleep onset | At 16 weeks after beginning study
  Assessed by an Actigraph 2 monitor

CONTACTS AND LOCATIONS:
Overall Officials: Alison Shea, MD, Principal Investigator — St. Joseph's Healthcare, McMaster University
Locations (1):
- St Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No